CLINICAL TRIAL: NCT03026777
Title: Preventing Cardiovascular collaPse With Administration of Fluid Resuscitation Before Endotracheal Intubation: The PrePARE Trial
Brief Title: Preventing Cardiovascular collaPse With Administration of Fluid Resuscitation Before Endotracheal Intubation
Acronym: PrePARE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center in New Orleans (Other)
Responsible Party: Principal Investigator, David Janz, Assistant Professor of Medicine, Louisiana State University Health Sciences Center in New Orleans
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Prepare
Record Dates: First submitted 2017-01-17; First posted 2017-01-20 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2020-12

CONDITIONS: Acute Respiratory Failure; Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Fluid Loading (Experimental): (1) 500 milliliters of an intravenous crystalloid solution of the operator's choosing will be (2) infused at any time after randomization and prior to the administration of procedural medications from (3) above the level of the central or peripheral intravenous or intraosseus access used and allowed to infuse by gravity and (4) stopped after 500 mL have infused. All intravenous infusions preceding the decision to perform endotracheal intubation will not be altered.
  Interventions: Drug: intravenous crystalloid fluid, 500 mL
- Usual Care (No Intervention): No intravenous fluids are started after the decision is made to perform endotracheal intubation. All intravenous infusions preceding the decision to perform endotracheal intubation will not be altered.

INTERVENTIONS:
Drug: intravenous crystalloid fluid, 500 mL
  Arms: Fluid Loading

SUMMARY:
Endotracheal intubation is common in the care of critically ill patients. Complications of airway management in this setting are frequently encountered and may be associated with an increased risk of death. The prevention of complications during urgent and emergent endotracheal intubation is a key focus for airway management research. Post-intubation hypotension (PIH), a common complication of endotracheal intubation in the critically ill, may be prevented by a bolus of intravenous fluid prior to the start of the procedure, but this approach has not been examined in a prospective trial. There are no randomized trials of intravenous fluid administration to prevent PIH in critically ill adults. The investigators propose a randomized trial of fluid loading to prevent PIH in critically ill adults.

DETAILED DESCRIPTION:
The investigators propose a randomized, parallel-group trial evaluating the impact of fluid loading to decrease cardiovascular collapse during and after endotracheal intubation in critically ill adults. Patients admitted to the study sites who are deemed by their clinical team to require intubation and fulfill inclusion criteria without meeting exclusion criteria will be enrolled and randomly assigned to intravenous fluid loading versus none. All other decisions regarding airway management will remain at the discretion of the treating provider. Data will be collected at the time of intubation and prospectively from the medical record in order to determine the effect of the assigned intervention on short- and long-term outcomes. All data are collected non-invasively and are already a part of clinical data obtained in usual ICU care at the bedside or in the medical record. No additional data will be collected that is not observed at the bedside or obtained from the medical record.

Study Population: The study population will be all critically ill adults for whom the clinical team has decided to perform endotracheal intubation using sedation with or without neuromuscular blockade. Patients will be excluded only if the operator feels: 1. Additional intravenous fluids in the form of fluid loading is absolutely indicated or contraindicated, or 2. The urgency of the intubation would make performing the study procedures unsafe. Patients will be included regardless of gender, race, weight or body mass index, initial oxygen saturation, anticipated grade of view, and other clinical factors.

Study Interventions:

Fluid Loading - (1) 500 milliliters of an intravenous crystalloid solution of the operator's choosing will be (2) infused at any time after randomization and prior to the administration of procedural medications from (3) above the level of the central or peripheral intravenous or intraosseus access used and allowed to infuse by gravity and (4) stopped after 500 mL have infused. All intravenous infusions preceding the decision to perform endotracheal intubation will not be altered.

No Fluid Loading - No intravenous fluids are started after the decision is made to perform endotracheal intubation. All intravenous infusions preceding the decision to perform endotracheal intubation will not be altered.

Primary Endpoint:

Cardiovascular collapse - a composite endpoint defined as one or more of the following:

* Death within 1 hour of intubation
* Cardiac arrest within 1 hour of intubation
* New systolic blood pressure < 65 mmHg between induction and 2 minutes after completion of intubation
* New or increased vasopressor receipt between induction and 2 minutes after completion of intubation

ELIGIBILITY:
Inclusion Criteria:

* Patient is admitted to participating study unit
* Planned procedure is endotracheal intubation and planned operator is a provider expected to routinely perform endotracheal intubation in the participating unit
* Administration of sedation with or without neuromuscular blockade is planned
* Age ≥ 18 years old

Exclusion Criteria:

* Operator believes fluid loading to be absolutely indicated or contraindicated for the safe care of the patient
* Urgency of intubation precludes safe performance of study procedures
* Pregnancy
* Prisoners
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 337 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Janz, MD, MSc, Study Chair — LSU School of Medicine New Orleans
Locations (7):
- United States (7):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Ochsner Medical Center, Jefferson, Louisiana
  - LSUHSC and University Medical Center, New Orleans, Louisiana
  - Lahey Medical Center, Burlington, Massachusetts
  - Lincoln Medical Center, The Bronx, New York
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Janz DR, Casey JD, Semler MW, Russell DW, Dargin J, Vonderhaar DJ, Dischert KM, West JR, Stempek S, Wozniak J, Caputo N, Heideman BE, Zouk AN, Gulati S, Stigler WS, Bentov I, Joffe AM, Rice TW; PrePARE Investigators; Pragmatic Critical Care Research Group. Effect of a fluid bolus on cardiovascular collapse among critically ill adults undergoing tracheal intubation (PrePARE): a randomised controlled trial. Lancet Respir Med. 2019 Dec;7(12):1039-1047. doi: 10.1016/S2213-2600(19)30246-2. Epub 2019 Oct 1. PMID 31585796

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluid Loading: (1) 500 milliliters of an intravenous crystalloid solution of the operator's choosing will be (2) infused at any time after randomization and prior to the administration of procedural medications from (3) above the level of the central or peripheral intravenous or intraosseus access used and allowed to infuse by gravity and (4) stopped after 500 mL have infused. All intravenous infusions preceding the decision to perform endotracheal intubation will not be altered.
  intravenous crystalloid fluid, 500 mL
Period: Overall Study
Arm/Group | Fluid Loading | Usual Care
Started | 168 | 169
Completed | 168 | 169
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All patients randomized were included in the baseline analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluid Loading | Usual Care | Total
Number analyzed (Participants) | 168 | 169 | 337
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [47 to 70] | 58 [46 to 68] | 60 [49 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 73 | 154
  Male | 87 | 96 | 183
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Race | 115 | 121 | 236
  Other | 53 | 48 | 101
Region of Enrollment [Number; unit: participants]
  United States | 168 | 169 | 337
Body-mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 27 [14 to 27] | 26 [22 to 32] | 26 [22 to 30]
Acute physiology and chronic health evaluation score [Median (Inter-Quartile Range); unit: units on a scale, range 0 to 71] — range 0 to 71, higher scores indicate a higher severity of illness
  units on a scale, range 0 to 71 | 21 [14 to 27] | 20 [16 to 27] | 20 [16 to 27]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Cardiovascular Collapse
Description: a composite endpoint defined as one or more of the following:
  * Death within 1 hour of intubation
  * Cardiac arrest within 1 hour of intubation
  * New systolic blood pressure < 65 mmHg between induction and 2 minutes after completion of intubation
  * New or increased vasopressor receipt between induction and 2 minutes after completion of intubation
Time Frame: 1 hour
Population: All patients randomized were included in the primary analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
Participants | 33 | 31

2. Secondary Outcome: In-hospital Mortality
Description: What was the patient's vital status at the time of hospital discharge
Time Frame: from date of randomization through study completion, an average of 28 days
Population: intention to treat
Measure: Count of Participants; unit: Participants
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
Participants | 48 | 59

3. Secondary Outcome: Ventilator-free Days
Description: Number of days alive and free of invasive ventilation in a 28-day period
Time Frame: from date of randomization through study completion, an average of 28 days
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
days | 20 [0 to 25] | 19 [0 to 25]

4. Secondary Outcome: ICU-free Days
Description: Number of days alive and outside of an ICU in a 28 day period
Time Frame: from date of randomization through study completion, an average of 28 days
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
days | 16 [0 to 24] | 14 [0 to 23]

5. Secondary Outcome: Lowest Arterial Oxygen Saturation
Description: Lowest arterial oxygen saturation between induction and 2 min after intubation
Time Frame: between induction and 2 minutes following procedure
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: percentage of hemoglobin
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
percentage of hemoglobin | 94 [84 to 99] | 95 [82 to 99]

6. Secondary Outcome: Number of Laryngoscopy Attempts
Description: Number of laryngoscopy attempts to achieve successful tracheal intubation
Time Frame: during procedure
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: attempts
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
attempts | 1 [1 to 1] | 1 [1 to 1]

7. Secondary Outcome: Lowest Systolic Blood Pressure
Description: Lowest systolic blood pressure between induction and 2 min after intubation
Time Frame: between induction and 2 minutes following procedure
Population: intention to treat
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | Fluid Loading | Usual Care
Number analyzed (Participants) | 168 | 169
mmHg | 119 [95 to 140] | 119 [94 to 141]

ADVERSE EVENTS:
Time Frame: 28 days after enrollment and randomization
Arm/Group | Fluid Loading | Usual Care
All-Cause Mortality (participants affected / at risk) | 48/168 | 59/169
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/169
Other Adverse Events (participants affected / at risk) | 0/168 | 0/169

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03026777/SAP_000.pdf
  • Study Protocol (2020-12-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT03026777/Prot_001.pdf